CLINICAL TRIAL: NCT06451224
Title: Attitudes of Prophylactic Antibiotic Utilization During Primary Total Hip and Knee Arthroplasty Among Egyptian Joint Replacement Surgeons
Brief Title: Egyptian Arthroplasty Surgeons' Antibiotics Usage Awareness
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed A. Khalifa, MD, FRCS, MSc, Assistant Professor, South Valley University
Other Study IDs: 04-2024-300439
Record Dates: First submitted 2024-05-23; First posted 2024-06-11 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Infections Joint Prosthetic
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — Online Questionnaire

SUMMARY:
Total hip arthroplasty (THA) and total knee arthroplasty (TKA) are procedures successfully applied to manage various end-stage chronic hip and knee diseases, such as osteoarthritis, rheumatoid arthritis, and femoral head avascular necrosis, as well as acute conditions, such as the neck of femur fractures, with excellent long-term functional outcomes. One of the devastating complications after such a procedure is periprosthetic joint infection (PJI). Various precautions are proposed to guard against such complications; one is the administration of perioperative antibiotics. However, injudicious or misuse of antibiotics could lead to the emergence of antimicrobial resistance, further complicating this matter. This is why various scientific and research organizations have proposed guidelines and a consensus for proper antibiotic use in perioperative THA and TKA surgery.

Antibiotic prophylaxis during primary THA and TKA can reduce the risk of PJI and surgical site infections. However, there is a lack of consensus on the optimal dosages and duration of prophylaxis, and guidelines vary among institutions. Alternatives such as extended oral antibiotic prophylaxis and different antibiotic regimens are being explored. International research is needed to establish best practices and determine the potential risks of antibiotic prophylaxis during primary THA and TKA. Unfortunately, the investigators are unaware of such guidelines proposed by any Egyptian health authority to guide and control the proper utilization of antibiotics during orthoapedic practice in general and joint replacement surgeries (THA and TKA) in particular.

DETAILED DESCRIPTION:
This study will be an Online-based questionnaire investigating surgeons' perspectives on antibiotics utilization during primary total hip and knee arthroplasty surgeries and investigate their thoughts about the necessity for developing local guidelines.

ELIGIBILITY:
Inclusion criteria:

All Egyptian registered members of the Egyptian Pelvis and Hip Society, practicing Egyptian joint replacement surgeons (performing surgeries as a leading surgeon) who are willing to participate

Exclusion criteria:

* Members not listed in the E-mail directory of the society
* Surgeons refusing to participate
* Young surgeons who are not practicing independently

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active practicing Egyptian joint replacement surgeons
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
To determine the type of antibiotics administration during primary total hip and knee arthroplasty | 2 months
  The type of antibiotics will be determined as follows: the name of the antibiotic (brand or generic), and if single or dual antibiotics are used. These will be presented as numbers and percentages.

SECONDARY OUTCOMES:
To determine the dose of antibiotics administered during primary total hip and knee arthroplasty | 2 months
  The dose of antibiotics will be determined as grams or milligrams. Furthermore, the number of doses will be reported
To determine the timing of antibiotics administration during primary total hip and knee arthroplasty | 2 months
  Regarding the timing, preoperative antibiotic administration will be reported in minutes
To determine the length of antibiotics administration during primary total hip and knee arthroplasty | 2 months
  the length of antibiotic administration postoperatively will be calculated in days.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abd El-Aal, MD, Study Chair — Assiut University
Locations (1):
- Assuit Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided